CLINICAL TRIAL: NCT05272280
Title: Ultrasound Guided External Oblique Intercostal (EOI) Block Versus Erector Spinae Plane Block (ESPB) for Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: US Guided EOI Block Versus ESPB for Postoperative Analgesia in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Magdy Mohammed Mahdy Sayed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABC-5-DE
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
Keywords: Cholecystectomy; EOI block; ESP block
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: triple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External oblique intercostal (EOI) block (Active Comparator)
  Interventions: Other: External oblique intercostal (EOI) block
- Erector spinae plane block (ESPB) (Active Comparator)
  Interventions: Other: Erector spinae plane block (ESPB)

INTERVENTIONS:
Other: External oblique intercostal (EOI) block — A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation at the sixth intercostal space in the anterior midaxillary line. A 21G 10 cm needle will be inserted using an in plane approach. The tip of the needle will be placed into the fascial plane on the deep aspect of the external oblique muscle. A volume of 20 mL of LA mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a mixture totaling 20 ml.) will be injected. The same procedure will be repeated for the opposite side.
  Arms: External oblique intercostal (EOI) block
Other: Erector spinae plane block (ESPB) — A high-frequency linear ultrasound probe will be placed in a longitudinal parasagittal orientation 2.5-3 cm lateral to the T9 spinous process. The erector spinae muscles will be identified superficial to the tip of the T9 transverse process. A 21G 10 cm needle will be inserted using an in plane approach. The tip of the needle will be placed into the fascial plane on the deep aspect of the erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting the erector spinae muscle off the bony shadow of the transverse process on ultrasonographic imaging. A volume of 20 mL of Local Anesthetic mixture (10 mL of bupivacaine 0.5%, 5 mL of lidocaine 2% and 5 mL of normal saline to make a mixture totaling 20 ml.) will be injected. The same procedure will be repeated for the opposite side.
  Arms: Erector spinae plane block (ESPB)

SUMMARY:
To compare the efficacy of USG-guided bilateral External oblique intercostal (EOI) block with Erector spinae plane block (ESPB) for post-operative analgesia after laparoscopic cholecystectomy with a hypothesis that both External oblique intercostal fascial plane block and Erector spinae plane block are effective in providing post-operative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years with a body mass index (BMI) of 18-35 kg/m2,
* patients with the American Society of Anesthesiologists (ASA) physical status I/II,
* Patients scheduled for elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Allergy to local anaesthetics,
* Infection at the site of injection,
* Coagulopathy,
* Chronic pain syndromes,
* Prolonged opioid medication,
* Patients who received any analgesic 24 h before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Nalbuphine consumption in mg equivalent to morphine dose. | 24 hours postoperatively
  mg

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) at rest and when coughing | at 1, 2,4 , 8, 16 and 24 hours postoperatively
  11-point scale where 0=no pain and 10=worst pain
Analgesic drug consumption other than nalbuphine | 24 hours postoperatively
  in mg
Heart Rate | Intraoperatively at 0, 5,10, 20, and 30 minutes. Then every 15 min thereafter till the end of surgery
  beats /min
Mean Arterial Pressure | Intraoperatively at 0, 5,10, 20, and 30 minutes. Then every 15 min thereafter till the end of surgery
  mmHg
Incidence of Postoperative nausea & vomiting (PONV) | 24 hours postoperatively
  Number of patients developing PONV
Shoulder pain | 24 hours postoperatively
  Number of patients developing Shoulder pain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Assiut, Asyut Governorate, Egypt,, Egypt